CLINICAL TRIAL: NCT00491244
Title: Pegylated Interferon Alfa-2a Plus Low Dose Ribavirin Versus Pegylated Interferon Alfa-2a Alone for Treatment-naïve Hemodialysis Patients With Chronic Hepatitis C
Brief Title: Pegylated Interferon Alfa-2a Plus Low Dose Ribavirin for Treatment-Naïve Hemodialysis Patients With Chronic Hepatitis C
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government); Department of Health, Executive Yuan, R.O.C. (Taiwan) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200703010M
Record Dates: First submitted 2007-06-23; First posted 2007-06-26 (Estimated); Results first posted 2013-12-13 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-01

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic hepatitis C; Hemodialysis; Interferon; Ribavirin
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peginterferon alfa-2a and ribavirin (Experimental): Pegylated interferon alfa-2a (Pegasys, F. Hoffman-LaRoche) 135 ug/week plus ribavirin (Copegus, F. Hoffman-LaRoche) 200 mg/day for 24 to 48 weeks (genotype 1: 48 weeks, genotype 2: 24 weeks)
  Interventions: Drug: Peginterferon alfa-2a and ribavirin
- Peginterferon alfa-2a (Experimental): Pegylated interferon alfa-2a (Pegasys, F. Hoffman-LaRoche) 135 ug/week for 24 to 48 weeks (genotype 1: 48 weeks, genotype 2: 24 weeks)
  Interventions: Drug: Peginterferon alfa-2a

INTERVENTIONS:
Drug: Peginterferon alfa-2a and ribavirin — Pegylated interferon alfa-2a (Pegasys, F. Hoffman-LaRoche) 135 ug/week plus ribavirin (Copegus, F. Hoffman-LaRoche) 200 mg/day for 24 to 48 weeks (genotype 1: 48 weeks, genotype 2: 24 weeks)
  Other Names: Pegylated interferon alfa-2a (Pegasys, F. Hoffman-LaRoche); Ribavirin (Copegus, F. Hoffman-LaRoche)
  Arms: Peginterferon alfa-2a and ribavirin
Drug: Peginterferon alfa-2a — Pegylated interferon alfa-2a (Pegasys, F. Hoffman-LaRoche) 135 ug/week for 24 to 48 weeks (genotype 1: 48 weeks, genotype 2: 24 weeks)
  Other Names: Pegylated interferon alfa-2a (Pegasys, F. Hoffman-LaRoche)
  Arms: Peginterferon alfa-2a

SUMMARY:
Chronic hepatitis C virus (HCV) infection is common in dialysis patients. Interferon (IFN)-based treatment for chronic hepatitis C has been the mainstay therapy in immunocompetent patients. In dialysis patients, treatment with conventional or pegylated interferon has also received much attention recently. Two meta-analyses evaluating the efficacy and safety of conventional IFN alfa monotherapy showed that the sustained virologic response (SVR) rates were 37% and 33%, respectively; and the corresponding dropout rates were 17% and 29.6%, respectively.The efficacy and safety of pegylated IFN alfa-2a and 2b in treating dialysis patients showed conflicting results, with a more favorable outcome of patients treated with pegylated IFN alfa-2a (135-180 μg/week: SVR 33-75%, well tolerated) than those treated with pegylated IFN alfa-2b (0.5-1.0 μg/week: SVR 12.5%, poorly tolerated. Currently, IFN-based therapy to treatment HCV infection should be initiated in dialysis stages, because the use of IFN in RT patients harbors high risks of acute graft rejection,and have low response rates under the concomitant use of immunosuppressive agents.

Ribavirin, which has been used in combination with IFN to treat chronic hepatitis C in the general patients and achieve a higher SVR rate than IFN monotherapy, is considered contraindicated in dialysis patients with chronic hepatitis C due to the risk of severe hemolytic anemia. However, some pilot studies evaluating combined conventional IFN alfa plus low dose ribavirin (170-300 mg/day) showed SVR rates of 17%-66% after 24-48 weeks of treatment. In addition, a recent study including 6 patients with combination of pegylated IFN alfa plus low dose ribavirin also showed a SVR rate of 50%. In this study, treatment with pegylated IFN alfa-2a plus low dose ribavirin achieved a higher SVR rate that that with pegylated IFN alfa-2b plus low dose ribavirin (100% vs. 25%).

Based on the long-term favorable outcome in dialysis patients who eradicate HCV, and the superior response of pegylated IFN alfa-2a plus low dose ribavirin to pegylated IFN alfa-2b plus low dose ribavirin in treating dialysis patients with chronic hepatitis C, the aim of the study is to evaluate the efficacy and safety of pegylated IFN alfa-2a plus low dose ribavirin versus pegylated interferon alfa-2a alone in treatment naïve dialysis patients with chronic hepatitis C.

DETAILED DESCRIPTION:
Chronic hepatitis C virus (HCV) infection is common in dialysis patients, with the reported prevalence varying from 3% to 80% worldwide. (1-3) Although these patients usually have mild symptoms and moderate elevation of alanine transaminase levels, recent international collaborative survey and prospective studies found that anti-HCV seropositivity and positive HCV RNA were risk factors for mortality and hepatocellular carcinoma (HCC). (4-7) Furthermore, progressive hepatic fibrosis, poor patient and graft survival were observer in dialysis patients with HCV infection who undergo renal transplantation (RT), suggesting immunosuppression following RT may worsen the course of hepatic fibrosis and renal graft function. (8-13) These lines of evidence indicate that HCV infection in the dialysis population is an important issue to be tackled.

Interferon (IFN)-based treatment for chronic hepatitis C has been the mainstay therapy in immunocompetent patients. In dialysis patients, treatment with conventional or pegylated interferon has also received much attention recently. Two meta-analyses evaluating the efficacy and safety of conventional IFN alfa monotherapy showed that the sustained virologic response (SVR) rates were 37% and 33%, respectively; and the corresponding dropout rates were 17% and 29.6%, respectively.(14,15) The efficacy and safety of pegylated IFN alfa-2a and 2b in treating dialysis patients showed conflicting results, with a more favorable outcome of patients treated with pegylated IFN alfa-2a (135-180 μg/week: SVR 33-75%, well tolerated) than those treated with pegylated IFN alfa-2b (0.5-1.0 μg/week: SVR 12.5%, poorly tolerated), (16-21) which may result from different pharmacokinetic profiles between these two pegylated IFNs. Currently, IFN-based therapy to treatment HCV infection should be initiated in dialysis stages, because the use of IFN in RT patients harbors high risks of acute graft rejection,(22,23) and have low response rates under the concomitant use of immunosuppressive agents. (24,25) Ribavirin, which has been used in combination with IFN to treat chronic hepatitis C in the general patients and achieve a higher SVR rate than IFN monotherapy, is considered contraindicated in dialysis patients with chronic hepatitis C due to the risk of severe hemolytic anemia. However, some pilot studies evaluating combined conventional IFN alfa plus low dose ribavirin (170-300 mg/day) showed SVR rates of 17%-66% after 24-48 weeks of treatment. (26-28) In addition, a recent study including 6 patients with combination of pegylated IFN alfa plus low dose ribavirin also showed a SVR rate of 50%. (29) In this study, treatment with pegylated IFN alfa-2a plus low dose ribavirin achieved a higher SVR rate that that with pegylated IFN alfa-2b plus low dose ribavirin (100% vs. 25%) Based on the long-term favorable outcome in dialysis patients who eradicate HCV, and the superior response of pegylated IFN alfa-2a plus low dose ribavirin to pegylated IFN alfa-2b plus low dose ribavirin in treating dialysis patients with chronic hepatitis C, the aim of the study is to evaluate the efficacy and safety of pegylated IFN alfa-2a plus low dose ribavirin versus pegylated interferon alfa-2a in treatment naïve dialysis patients with chronic hepatitis C.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old
* Creatinine clearance (Ccr) < 15 ml/min/1.73 m2
* Anti-HCV (Abbott HCV EIA 3.0, Abbott Diagnostic, Chicago, IL) positive > 6 months
* Detectable serum quantitative HCV-RNA (Cobas Taqman HCV test, version 2, Roche Diagnostics) with a dynamic range of 25-391000000 IU/ml

Exclusion Criteria:

* Receiving interferon-based therapy for chronic hepatitis C
* Severe anemia (hemoglobin < 10 g/dL) or hemoglobinopathy
* Neutropenia (neutrophil count, <1,500/mm3)
* Thrombocytopenia (platelet <90,000/ mm3)
* Co-infection with HBV or HIV
* Chronic alcohol abuse (daily consumption > 20 g/day)
* Autoimmune liver disease
* Decompensated liver disease (Child classification B or C)
* Neoplastic disease
* An organ transplant
* Immunosuppressive therapy
* Poorly controlled autoimmune diseases, pulmonary diseases, cardiac diseases, psychiatric diseases, neurological diseases, diabetes mellitus
* Evidence of drug abuse
* Unwilling to have contraception

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 377 (Actual)
Dates: Start 2007-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Hua Liu, MD, Study Chair — Department of Internal Medicine, National Taiwan Universitys Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Fabrizi F, Poordad FF, Martin P. Hepatitis C infection and the patient with end-stage renal disease. Hepatology. 2002 Jul;36(1):3-10. doi: 10.1053/jhep.2002.34613. PMID 12085342
- [Background] Kao JH, Huang CH, Chen W, Tsai TJ, Lee SH, Hung KY, Chen DS. GB virus C infection in hemodialysis patients: molecular evidence for nosocomial transmission. J Infect Dis. 1999 Jul;180(1):191-4. doi: 10.1086/314850. PMID 10353878
- [Background] Hou CH, Chen WY, Kao JH, Chen DS, Yang Y, Chen JJ, Lee SH, Wu DJ, Yang SC. Intrafamilial transmission of hepatitis C virus in hemodialysis patients. J Med Virol. 1995 Apr;45(4):381-5. doi: 10.1002/jmv.1890450405. PMID 7545208
- [Background] Maisonneuve P, Agodoa L, Gellert R, Stewart JH, Buccianti G, Lowenfels AB, Wolfe RA, Jones E, Disney AP, Briggs D, McCredie M, Boyle P. Cancer in patients on dialysis for end-stage renal disease: an international collaborative study. Lancet. 1999 Jul 10;354(9173):93-9. doi: 10.1016/s0140-6736(99)06154-1. PMID 10408483
- [Background] Nakayama E, Akiba T, Marumo F, Sato C. Prognosis of anti-hepatitis C virus antibody-positive patients on regular hemodialysis therapy. J Am Soc Nephrol. 2000 Oct;11(10):1896-1902. doi: 10.1681/ASN.V11101896. PMID 11004221
- [Background] Stehman-Breen CO, Emerson S, Gretch D, Johnson RJ. Risk of death among chronic dialysis patients infected with hepatitis C virus. Am J Kidney Dis. 1998 Oct;32(4):629-34. doi: 10.1016/s0272-6386(98)70027-7. PMID 9774125
- [Background] Pereira BJ, Natov SN, Bouthot BA, Murthy BV, Ruthazer R, Schmid CH, Levey AS. Effects of hepatitis C infection and renal transplantation on survival in end-stage renal disease. The New England Organ Bank Hepatitis C Study Group. Kidney Int. 1998 May;53(5):1374-81. doi: 10.1046/j.1523-1755.1998.00883.x. PMID 9573555
- [Background] Mathurin P, Mouquet C, Poynard T, Sylla C, Benalia H, Fretz C, Thibault V, Cadranel JF, Bernard B, Opolon P, Coriat P, Bitker MO. Impact of hepatitis B and C virus on kidney transplantation outcome. Hepatology. 1999 Jan;29(1):257-63. doi: 10.1002/hep.510290123. PMID 9862875
- [Background] Legendre C, Garrigue V, Le Bihan C, Mamzer-Bruneel MF, Chaix ML, Landais P, Kreis H, Pol S. Harmful long-term impact of hepatitis C virus infection in kidney transplant recipients. Transplantation. 1998 Mar 15;65(5):667-70. doi: 10.1097/00007890-199803150-00011. PMID 9521201
- [Background] Vosnides GG. Hepatitis C in renal transplantation. Kidney Int. 1997 Sep;52(3):843-61. doi: 10.1038/ki.1997.403. No abstract available. PMID 9291208
- [Background] Izopet J, Rostaing L, Sandres K, Cisterne JM, Pasquier C, Rumeau JL, Duffaut M, Durand D, Puel J. Longitudinal analysis of hepatitis C virus replication and liver fibrosis progression in renal transplant recipients. J Infect Dis. 2000 Mar;181(3):852-8. doi: 10.1086/315355. PMID 10720504
- [Background] Zylberberg H, Nalpas B, Carnot F, Skhiri H, Fontaine H, Legendre C, Kreis H, Brechot C, Pol S. Severe evolution of chronic hepatitis C in renal transplantation: a case control study. Nephrol Dial Transplant. 2002 Jan;17(1):129-33. doi: 10.1093/ndt/17.1.129. PMID 11773476
- [Background] Fabrizi F, Dulai G, Dixit V, Bunnapradist S, Martin P. Meta-analysis: interferon for the treatment of chronic hepatitis C in dialysis patients. Aliment Pharmacol Ther. 2003 Dec;18(11-12):1071-81. doi: 10.1046/j.1365-2036.2003.01780.x. PMID 14653826
- [Background] Russo MW, Goldsweig CD, Jacobson IM, Brown RS Jr. Interferon monotherapy for dialysis patients with chronic hepatitis C: an analysis of the literature on efficacy and safety. Am J Gastroenterol. 2003 Jul;98(7):1610-5. doi: 10.1111/j.1572-0241.2003.07526.x. PMID 12873587
- [Background] Kokoglu OF, Ucmak H, Hosoglu S, Cetinkaya A, Kantarceken B, Buyukbese MA, Isik IO. Efficacy and tolerability of pegylated-interferon alpha-2a in hemodialysis patients with chronic hepatitis C. J Gastroenterol Hepatol. 2006 Mar;21(3):575-80. doi: 10.1111/j.1440-1746.2005.04008.x. PMID 16638102
- [Background] Sporea I, Popescu A, Sirli R, Golea O, Totolici C, Danila M, Vernic C. Pegylated-interferon alpha 2a treatment for chronic hepatitis C in patients on chronic haemodialysis. World J Gastroenterol. 2006 Jul 14;12(26):4191-4. doi: 10.3748/wjg.v12.i26.4191. PMID 16830372
- [Background] Chan TM, Ho SK, Tang CS, Tse KC, Lam MF, Lai KN, Yung S. Pilot study of pegylated interferon-alpha 2a in dialysis patients with chronic hepatitis C virus infection. Nephrology (Carlton). 2007 Feb;12(1):11-7. doi: 10.1111/j.1440-1797.2006.00662.x. PMID 17295655
- [Background] Russo MW, Ghalib R, Sigal S, Joshi V. Randomized trial of pegylated interferon alpha-2b monotherapy in haemodialysis patients with chronic hepatitis C. Nephrol Dial Transplant. 2006 Feb;21(2):437-43. doi: 10.1093/ndt/gfi231. Epub 2005 Oct 18. PMID 16234288
- [Background] Annicchiarico BE, Siciliano M. Pegylated interferon-alpha 2b monotherapy for haemodialysis patients with chronic hepatitis C. Aliment Pharmacol Ther. 2004 Jul 1;20(1):123-4; author reply 124. doi: 10.1111/j.1365-2036.2004.01954.x. No abstract available. PMID 15225179
- [Background] Potthoff A, Wiegand J, Luth JB, Wedemeyer H, Manns MP, Tillmann HL. Superiority of standard interferon-alpha2b compared to pegylated interferon-alpha2b (12 kDa) in a hemodialysis patient with chronic hepatitis C? Clin Nephrol. 2005 Mar;63(3):232-5. doi: 10.5414/cnp63232. PMID 15786827
- [Background] Magnone M, Holley JL, Shapiro R, Scantlebury V, McCauley J, Jordan M, Vivas C, Starzl T, Johnson JP. Interferon-alpha-induced acute renal allograft rejection. Transplantation. 1995 Apr 15;59(7):1068-70. doi: 10.1097/00007890-199504150-00030. No abstract available. PMID 7709447
- [Background] Morales JM. Hepatitis C virus infection and renal disease after renal transplantation. Transplant Proc. 2004 Apr;36(3):760-2. doi: 10.1016/j.transproceed.2004.03.041. PMID 15110654
- [Background] Rostaing L, Izopet J, Baron E, Duffaut M, Puel J, Durand D. Treatment of chronic hepatitis C with recombinant alpha 2b interferon in kidney transplant recipients: preliminary results and side effects. Transplant Proc. 1995 Feb;27(1):948-50. No abstract available. PMID 7879242
- [Background] Casanovas-Taltavull T, Baliellas C, Benasco C, Serrano TT, Casanova A, Perez JL, Guerrero L, Gonzalez MT, Andres E, Gil-Vernet S, Casais LA. Efficacy of interferon for chronic hepatitis C virus-related hepatitis in kidney transplant candidates on hemodialysis: results after transplantation. Am J Gastroenterol. 2001 Apr;96(4):1170-7. doi: 10.1111/j.1572-0241.2001.03697.x. PMID 11316166
- [Background] Mousa DH, Abdalla AH, Al-Shoail G, Al-Sulaiman MH, Al-Hawas FA, Al-Khader AA. Alpha-interferon with ribavirin in the treatment of hemodialysis patients with hepatitis C. Transplant Proc. 2004 Jul-Aug;36(6):1831-4. doi: 10.1016/j.transproceed.2004.07.025. PMID 15350490
- [Background] Bruchfeld A, Stahle L, Andersson J, Schvarcz R. Ribavirin treatment in dialysis patients with chronic hepatitis C virus infection--a pilot study. J Viral Hepat. 2001 Jul;8(4):287-92. doi: 10.1046/j.1365-2893.2001.00300.x. PMID 11454181
- [Background] Bruchfeld A, Stahle L, Andersson J, Schvarcz R. Interferon and ribavirin therapy in dialysis patients with chronic hepatitis C. Nephrol Dial Transplant. 2001 Aug;16(8):1729. doi: 10.1093/ndt/16.8.1729. No abstract available. PMID 11477195
- [Background] Bruchfeld A, Lindahl K, Reichard O, Carlsson T, Schvarcz R. Pegylated interferon and ribavirin treatment for hepatitis C in haemodialysis patients. J Viral Hepat. 2006 May;13(5):316-21. doi: 10.1111/j.1365-2893.2005.00680.x. PMID 16637862
- [Derived] Prabhu AR, Rao IR, Nagaraju SP, Rajwar E, Venkatesh BT, Nair N S, Pai G, Reddy NP, Suvarna D. Interventions for dialysis patients with hepatitis C virus (HCV) infection. Cochrane Database Syst Rev. 2023 Apr 25;4(4):CD007003. doi: 10.1002/14651858.CD007003.pub3. PMID 37096802
- [Derived] Liu CH, Liu CJ, Huang CF, Lin JW, Dai CY, Liang CC, Huang JF, Hung PH, Tsai HB, Tsai MK, Lee CY, Chen SI, Yang SS, Su TH, Yang HC, Chen PJ, Chen DS, Chuang WL, Yu ML, Kao JH. Peginterferon alfa-2a with or without low-dose ribavirin for treatment-naive patients with hepatitis C virus genotype 2 receiving haemodialysis: a randomised trial. Gut. 2015 Feb;64(2):303-11. doi: 10.1136/gutjnl-2014-307080. Epub 2014 Apr 19. PMID 24747867
- [Derived] Liu CH, Huang CF, Liu CJ, Dai CY, Liang CC, Huang JF, Hung PH, Tsai HB, Tsai MK, Chen SI, Lin JW, Yang SS, Su TH, Yang HC, Chen PJ, Chen DS, Chuang WL, Yu ML, Kao JH. Pegylated interferon-alpha2a with or without low-dose ribavirin for treatment-naive patients with hepatitis C virus genotype 1 receiving hemodialysis: a randomized trial. Ann Intern Med. 2013 Dec 3;159(11):729-38. doi: 10.7326/0003-4819-159-11-201312030-00005. PMID 24297189

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from 1 June, 2007 to 9 May, 2012 Location: 8 academic centers in Taiwan
Groups:
- Peginterferon and Ribavirin: Pegylated interferon alfa-2a (Pegasys, F. Hoffman-LaRoche) 135 ug/week plus ribavirin (Copegus, F. Hoffman-LaRoche) 200 mg/day for 24 to 48 weeks (genotype 1: 48 weeks, genotype 2: 24 weeks)
- Peginterferon: Pegylated interferon alfa-2a (Pegasys, F. Hoffman-LaRoche) 135 ug/week for 24 to 48 weeks (genotype 1: 48 weeks, genotype 2: 24 weeks)
Period: Overall Study
Arm/Group | Peginterferon and Ribavirin | Peginterferon
Started | 189 | 188
Completed | 162 | 168
Not Completed | 27 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peginterferon and Ribavirin | Peginterferon | Total
Number analyzed (Participants) | 189 | 188 | 377
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 189 | 188 | 377
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (10) | 51 (11) | 51 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 76 | 152
  Male | 113 | 112 | 225
Region of Enrollment [Number; unit: participants]
  Taiwan | 189 | 188 | 377

OUTCOME MEASURES:

1. Primary Outcome: Sustained Virologic Response (SVR)Rate
Time Frame: 1.5 year
Population: All participants were analyzed if they received at least one dose of the study medication
Measure: Number; unit: participants
Arm/Group | Peginterferon and Ribavirin | Peginterferon
Number analyzed (Participants) | 189 | 188
participants | 130 | 72
Statistical Analysis 1: Comparison: Peginterferon and Ribavirin; Test type: Superiority or Other; p < 0.001, Chi-squared; Risk Ratio (RR) = 1.80, 95% CI 2-sided [1.46 to 2.21]

2. Secondary Outcome: Adverse Event (AE)-Related Withdrawal Rate
Time Frame: 1.5 year
Population: All patients were analyzed if they received at least one dose of the study medication; monitoring the events until the last visit
Measure: Number; unit: participants
Arm/Group | Peginterferon and Ribavirin | Peginterferon
Number analyzed (Participants) | 189 | 188
participants
  Advese event related withdrawal rate | 12 | 7
  Non withdrawal | 177 | 171
Statistical Analysis 1: Comparison: Peginterferon and Ribavirin; Test type: Superiority or Other; p = 0.35, Chi-squared; Risk Ratio (RR) = 1.61, 95% CI 2-sided [0.65 to 4.01]

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Peginterferon and Ribavirin | Peginterferon
Serious Adverse Events (participants affected / at risk) | 8/189 | 7/188
Other Adverse Events (participants affected / at risk) | 170/189 | 154/188
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peginterferon and Ribavirin (N=189) | Peginterferon (N=188)
Cholangitis (Infections and infestations) | 0 (0) | 1 (1)
Intractable diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1)
Peptic ulcer bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 3 (3)
Postural dizziness (Cardiac disorders) | 2 (2) | 0 (0)
Salmonella gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Stevens-Johnson sybdrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peginterferon and Ribavirin (N=189) | Peginterferon (N=188)
Flu-like syndrome (Immune system disorders) | 47 (47) | 50 (50)
Fatigue (Nervous system disorders) | 106 (106) | 97 (97)
Headache (Nervous system disorders) | 51 (51) | 48 (48)
Insomnia (Nervous system disorders) | 62 (62) | 66 (66)
Irritability (Psychiatric disorders) | 21 (21) | 19 (19)
Depression (Psychiatric disorders) | 25 (25) | 23 (23)
Anorexia (Gastrointestinal disorders) | 44 (44) | 38 (38)
Diarrhea (Gastrointestinal disorders) | 22 (22) | 20 (20)
Constipation (Gastrointestinal disorders) | 16 (16) | 15 (15)
Cough (Respiratory, thoracic and mediastinal disorders) | 26 (26) | 10 (10)
Dermatitis (Skin and subcutaneous tissue disorders) | 43 (43) | 38 (38)
Injection site reaction (Skin and subcutaneous tissue disorders) | 27 (27) | 27 (27)
Hair loss (Skin and subcutaneous tissue disorders) | 47 (47) | 43 (43)
Anemia (Blood and lymphatic system disorders) | 134 (134) | 13 (13) — Hemoglobin level < 8.5 g/dL
Neutropenia (Blood and lymphatic system disorders) | 30 (30) | 26 (26) — Absolute neutrophil count < 750 x 10^9 cells/L
Thrombocytopenia (Blood and lymphatic system disorders) | 19 (19) | 21 (21) — Platelet count < 50 x 10^9 cells/L

LIMITATIONS AND CAVEATS:
1. Open-label trial
2. Results may not be generalizable to peritoneal dialysis patients
3. Higher percentages of favorable IL28B genotypes
4. Secondary endpoint may not be powered to detect the differences

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No